CLINICAL TRIAL: NCT02783404
Title: An Oral Amoxicillin-Clavulanate Regimen to Prevent Bacteremia Following
Brief Title: An Oral Amoxicillin-Clavulanate Regimen to Prevent Bacteremia Following Dental Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Significant results (no control neither amoxicillin new arms needed)
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Pedro DIz DIos, MD, DDS, PhD, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Univ of Santiago de Compostela
Record Dates: First submitted 2016-05-22; First posted 2016-05-26 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Bacteraemia; Endocarditis
Keywords: bacteraemia; endocarditis; antibiotic prophylaxis; dentistry
MeSH Terms: conditions — Toxemia; Endocarditis | interventions — Amoxicillin; Drugs, Generic; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Receiving no prophylaxis
- Amoxicillin (Active Comparator): Receiving 2 gr oral Amoxicillin before any dental manipulation and following endotracheal intubation
  Intervention: Drug: Amoxicillin
  Interventions: Drug: Amoxicillin
- Amoxicillin-Potassium Clavulanate (Experimental): Receiving 2gr/125 mg oral Amoxicillin-Potassium Clavulanate before any dental manipulation and following endotracheal intubation
  Intervention: Drug: Amoxicillin-Potassium Clavulanate
  Interventions: Drug: Amoxicillin-Potassium Clavulanate

INTERVENTIONS:
Drug: Amoxicillin — Receiving 2 gr oral Amoxicillin before dental any manipulation and following endotracheal intubation
  Other Names: Amoxicillin (generic drug)
  Arms: Amoxicillin
Drug: Amoxicillin-Potassium Clavulanate — Receiving 2 gr/125 mg oral Amoxicillin-Potassium Clavulanate before any dental manipulation and following endotracheal intubation
  Intervention: Drug: Amoxicillin-Potassium Clavulanate
  Other Names: Amoxicillin-Potassium Clavulanate (generic drug)
  Arms: Amoxicillin-Potassium Clavulanate

SUMMARY:
Although controversy exists regarding the efficacy of antibiotic prophylaxis for patients at risk of infective endocarditis, expert committees continue to publish recommendations for antibiotic prophylactic regimens. Recently, the investigators have evaluated the efficacy of the intravenous administration of 1000/200 mg of amoxicillin/clavulanate for the prevention of bacteraemia following dental extractions. The results of this study suggest that is highly effective, and that it might be considered a first-line choice for patients at high-risk for infective endocarditis who undergo dental procedures and for whom antimicrobial prophylaxis is recommended. This new project aims to evaluate the effectiveness of oral amoxicillin/clavulanate in preventing post-dental extraction bloodstream infection.

DETAILED DESCRIPTION:
PURPOSE: Despite the controversy about the risk of developing bacterial endocarditis of oral origin, numerous Expert Committees in different countries continue to publish prophylactic regimens. To date, the literature is unclear about the role of antimicrobial prophylaxis in the prevention of bacteremia following dental procedures. The aim of this study is to evaluate the efficacy of prophylactic dosage with oral amoxicillin-clavulanate (AMX-CLV) in the prevention of bacteremia following dental extractions.

SELECTION OF THE STUDY GROUP AND STUDY DESIGN: The study group will comprise patients who, for behavioral reasons (autism, learning disabilities, phobias, etc.), will undergo dental extractions under general anesthesia in the Santiago de Compostela University Hospital (Santiago de Compostela, Spain). The following exclusion criteria will be applied: age under 18 years; body weight under 40 kg; receipt of antibiotics in the previous 3 months; routine use of oral antiseptics; a history of allergy or intolerance to AMX or CLV; any type of congenital or acquired immunodeficiency; or any known risk factor for bacterial endocarditis. By applying these criteria, 150 patients will be selected and will be randomly distributed into 3 study groups: control group (receiving no prophylaxis), AMX-CLV group (receiving 2 g/125 mg oral AMX-CLV), and AMX group (receiving 2 g oral AMX).

COLLECTION OF SAMPLES FOR BLOOD CULTURE: To determine the prevalence of bacteremia, a peripheral venous blood sample (10 ml) will be drawn from each patient at the baseline (before any dental manipulation but after nasotracheal intubation) and 30 s, 15 min, and 1 h after the final dental extraction. Samples will be inoculated in BACTEC plus (Becton Dickinson and Company, Sparks, MD) aerobic and anaerobic blood culture bottles, and will be processed in the Bactec 9240 (Becton Dickinson).

MICROBIOLOGICAL ANALYSIS OF BLOOD CULTURES: A Gram stain will be performed on each positive blood culture. The positive blood cultures in the aerobic media will be subcultured on blood agar and chocolate agar in an atmosphere of 5 to 10% carbon monoxide and on MacConkey agar under aerobic conditions. The same protocol will be used for the positive blood cultures in the anaerobic media, with subculture on Schaedler agar and incubation in an anaerobic atmosphere. The bacteria isolated will be identified by using the battery of biochemical tests provided with the Vitek system for Gram-positive bacteria, Neisseria spp., Haemophilus spp., and obligate anaerobic bacteria. The viridans group streptococci will be classified into five groups, the Streptococcus mitis, S. anginosus, S. salivarius, S. mutans, and S. bovis groups, by applying the Ruoff criteria. Facklam's criteria will be used to identify unusual Streptococcus spp. and other gram-positive cocci in chains.

The subculture and further identification of the isolated bacteria will be performed by conventional microbiological techniques. The collection, handling, and transport of the blood samples for blood culture will be performed according to the recommendations of the Spanish Society of Infectious Diseases and Clinical Microbiology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have at least 10 teeth
* Subjects must have the need for a dental extraction under general anesthesia (for behavioral reasons)
* Subjects will be recruited regardless of the extent and severity of their dental and/or periodontal disease

Exclusion Criteria:

* Age under 18 years
* Body weight under 40 kg
* Receipt of antibiotics in the previous 3 months
* Routine use of oral antiseptics
* A history of allergy or intolerance to amoxicillin
* A history of allergy or intolerance to chlorhexidine
* A history of allergy or intolerance to amoxicillin-clavulanate
* Any type of congenital or acquired immunodeficiency
* Any known risk factor for bacterial endocarditis
* Any known risk factor for prolonged bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Bacteremia in participants receiving a prophylactic dosage with oral amoxicillin-clavulanate | Changes from baseline in prevalence of bacteremia at 30 seconds, 15 minutes and 1 hour after the final dent
  Positive cultures

SECONDARY OUTCOMES:
Bacteremia in participants receiving a prophylactic dosage with oral amoxicillin | Changes from baseline in prevalence of bacteremia at 30 seconds, 15 minutes and 1 hour after the final dental extraction
  Positive cultures
Bacteremia in participants receiving no prophylaxis | Changes from baseline in prevalence of bacteremia at 30 seconds, 15 minutes and 1 hour after the final dental extraction
  Positive cultures

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Diz, MD, DDS, PhD, Principal Investigator — Santiago de Compostela University
Locations (2):
- Spain (2):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Santiago de Compostela University Hospital, Santiago de Compostela, Coruña

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available on request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: By the end of the study (for 1 year)
Access Criteria: On request

REFERENCES:
- [Background] Diz Dios P. Infective endocarditis prophylaxis. Oral Dis. 2014 May;20(4):325-8. doi: 10.1111/odi.12221. Epub 2014 Jan 13. PMID 24373017
- [Result] Valdes C, Tomas I, Alvarez M, Limeres J, Medina J, Diz P. The incidence of bacteraemia associated with tracheal intubation. Anaesthesia. 2008 Jun;63(6):588-92. doi: 10.1111/j.1365-2044.2008.05449.x. PMID 18477269
- [Result] Pineiro A, Tomas I, Blanco J, Alvarez M, Seoane J, Diz P. Bacteraemia following dental implants' placement. Clin Oral Implants Res. 2010 Sep;21(9):913-8. doi: 10.1111/j.1600-0501.2010.01928.x. PMID 20701619
- [Result] Diz Dios P, Tomas Carmona I, Limeres Posse J, Medina Henriquez J, Fernandez Feijoo J, Alvarez Fernandez M. Comparative efficacies of amoxicillin, clindamycin, and moxifloxacin in prevention of bacteremia following dental extractions. Antimicrob Agents Chemother. 2006 Sep;50(9):2996-3002. doi: 10.1128/AAC.01550-05. PMID 16940094
- [Result] Limeres Posse J, Alvarez Fernandez M, Fernandez Feijoo J, Medina Henriquez J, Lockhart PB, Chu VH, Diz Dios P. Intravenous amoxicillin/clavulanate for the prevention of bacteraemia following dental procedures: a randomized clinical trial. J Antimicrob Chemother. 2016 Jul;71(7):2022-30. doi: 10.1093/jac/dkw081. Epub 2016 Mar 29. PMID 27029851